CLINICAL TRIAL: NCT01212484
Title: Carbidopa for the Treatment of Nausea and Vomiting in Familial Dysautonomia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 09-0011
Record Dates: First submitted 2010-09-13; First posted 2010-09-30 (Estimated); Results first posted 2016-03-28 (Estimated); Last update posted 2016-03-28 (Estimated); Status verified 2016-03

CONDITIONS: Familial Dysautonomia
MeSH Terms: conditions — Dysautonomia, Familial | interventions — Carbidopa

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (first), Carbidopa (second) (Experimental): Crossover design Placebo first followed by carbidopa
  Interventions: Drug: Carbidopa; Drug: Placebo
- Carbidopa (first), Placebo (second) (Experimental): Crossover design carbidopa first followed by placebo
  Interventions: Drug: Carbidopa; Drug: Placebo

INTERVENTIONS:
Drug: Carbidopa — The trial will be divided into two consecutive, but independent parts. Phase 1, will address the safety and tolerability of carbidopa in patients with FD using an open-label dose titration phase followed by 4-weeks of open-label treatment. Phase 2, will address the efficacy of carbidopa for the treatment of nausea in patients with FD using a randomized, placebo controlled, double blind, 4-week cross over design.
  Other Names: Lodosyn
Drug: Placebo — The trial will be divided into two consecutive, but independent parts. Phase 1, will address the safety and tolerability of carbidopa in patients with FD using an open-label dose titration phase followed by 4-weeks of open-label treatment. Phase 2, will address the efficacy of carbidopa for the treatment of nausea in patients with FD using a randomized, placebo controlled, double blind, 4-week cross over design.

SUMMARY:
This is a pilot clinical trial of carbidopa to treat disabling attacks of nausea and vomiting in patients with familial dysautonomia (FD, also known as Riley Day syndrome or hereditary sensory and autonomic neuropathy type III). FD is a rare autosomal recessive disease in which the growth and development of selective nerves is impaired. Patients with FD suffer recurrent uncontrollable nausea and vomiting crises accompanied by skin flushing, tachycardia and arterial hypertension. Current treatments of nausea are ineffective or have intolerable side sides. Our long-term goal is to treat nausea effectively and without side effects, a therapeutic intervention that would markedly improve the quality of life of patients with FD.

The investigators have recently found that resting plasma dopamine levels are high in patients with FD and increase up to 40-fold during nausea and vomiting attacks. This led us to postulate that stimulation of dopamine receptors in the chemoreceptor trigger zone of the brainstem is the likely mechanism of vomiting.

Carbidopa is a reversible competitive inhibitor of aromatic L-amino acid decarboxylase (also known as dopa-decarboxylase) that cannot cross the blood brain barrier. It has been used successfully for many years to block the extracerebral synthesis of dopamine and avoid nausea and vomiting in patients with Parkinson's disease taking levodopa. The investigators reasoned that carbidopa could have a similar antiemetic effect in patients with FD.

The investigators propose to conduct a pilot trial to assess the safety, tolerability and efficacy of carbidopa for the treatment of nausea in patients with FD. The pilot trial will recruit 25 patients with FD who complain of severe nausea that affects their quality of life. The trial will be divided into two consecutive, but independent parts. Part 1, will address the safety and tolerability of carbidopa in patients with FD using an open-label dose titration phase followed by 4-weeks of open-label treatment. Part 2, will address the efficacy of carbidopa for the treatment of nausea in patients with FD using a randomized, placebo controlled, double blind, 4-week cross over design.

The investigators hope to demonstrate that carbidopa is a safe, well-tolerated drug that blocks the peripheral formation of dopamine and thus prevents dopamine-induced nausea and vomiting attacks in patients with FD.

DETAILED DESCRIPTION:
Patients with familial dysautonomia (FD), also called Riley Day syndrome or hereditary sensory and autonomic neuropathy type III, suffer recurrent attacks of uncontrollable nausea and vomiting that can last several hours or days and are severely disabling. Hypertension, tachycardia and skin blotching frequently accompany these attacks. Our long-term objective is to develop an effective treatment for nausea and vomiting in patients with FD.

In preliminary studies we found that plasma levels of dopamine were very high during attacks. Stimulation of dopamine receptors in the chemoreceptor trigger zone in the brainstem is a well-known cause of nausea and vomiting. The investigators postulate that acute increases in circulating dopamine levels are the cause of paroxysmal nausea and vomiting in FD.

Dopamine is synthesized by decarboxylation of the aminoacid L-dihydroxyphenylserine (L-DOPA) by the enzyme aromatic L-aminoacid decarboxylase, also known as DOPA decarboxylase. Patients with Parkinson's disease suffer nausea and vomiting when they receive treatment with L-DOPA. However, when L-DOPA is administered together with carbidopa, a reversible competitive inhibitor of DOPA decarboxylase that does not cross the blood brain barrier, nausea and vomiting are prevented. The investigators hypothesize that by blocking the conversion of DOPA to dopamine and thus preventing its increase in plasma, treatment with carbidopa will decrease nausea and vomiting in patients with FD.

Although carbidopa has been used for many years in patients with Parkinson's disease, it has never been used in patients with FD. The first specific aim of this proposal is to assess the safety and tolerability of carbidopa in patients with FD.

The second specific aim of this proposal is to determine whether blocking the peripheral synthesis of dopamine with carbidopa will improve recurrent nausea in patients with FD.

ELIGIBILITY:
Inclusion Criteria:

* Male of female patients aged 12 and older
* Confirmed diagnosis of familial dysautonomia by genetic testing.
* Symptoms of severe nausea
* Written informed consent or ascent to participate in the pilot trial and understanding that they can withdraw consent at anytime without affecting their future care.
* Ability to comply with the requirements of the study procedures, including taking blood pressure measurements at home.

Exclusion Criteria:

* Patients taking metroclopromide, domperidone, risperidone or other dopamine blockers
* Patients taking MAO-inhibitors
* Patients taking tricyclic antidepressants
* Patients taking neuroleptic drugs (haloperidol and chlorpromazine)
* Patients with a known hypersensitivity to any component of this drug.
* Patients with atrial fibrillation, angina or an electrocardiogram documenting significant abnormality that may jeopardize the patient's health.
* Patients with significant pulmonary, liver, renal (creatinine >2.0 mg/ml) or cardiac illness
* Patients who are unable to clearly identify and rate their symptoms of nausea.
* Women who are pregnant or lactating
* Patients who have a significant abnormality on clinical examination that may, in

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-12; Primary Completion 2012-02 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Horacio C Kaufmann, M.D., Principal Investigator — NYU Langone Health

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients were recruited at the NYU medical center's Dysautonomia Center.
Pre-assignment Details: Patients with FD that complain of severe nausea will be screened.
Groups:
- Placebo (First), Carbidopa (Second): Subjects will be given placebo first (4 weeks), followed by carbidopa (4 weeks).
- Carbidopa (First), Placebo (Second): Subjects will be given Carbidopa for a 4 week period followed by placebo for a 4 week period.
Period: Carbidopa Titration Period (4 Weeks)
Arm/Group | Placebo (First), Carbidopa (Second) | Carbidopa (First), Placebo (Second)
Started | 6 | 6
Completed | 5 | 6
Not Completed | 1 | 0
Period: First Intervention (4 Weeks)
Arm/Group | Placebo (First), Carbidopa (Second) | Carbidopa (First), Placebo (Second)
Started | 5 | 6
Completed | 5 | 4
Not Completed | 0 | 2
Period: Second Intervention (4 Weeks)
Arm/Group | Placebo (First), Carbidopa (Second) | Carbidopa (First), Placebo (Second)
Started | 5 | 4
Completed | 5 | 3
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Arm/Group | All Study Subjects
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8
  Between 18 and 65 years | 4
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.5 (6.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 8

OUTCOME MEASURES:

1. Primary Outcome: Composite Daily Score
Description: Daily scores were reported on a modified version of the Rhodes Index of Nausea, Vomiting and Retching, which included all 5 items relating to nausea and retching. Items addressing vomiting/throwing up were omitted, as all participants had antireflux surgery that prevented vomiting (Nissen fundoplication). Retching distress, nausea distress, number of nausea episodes per day, number of retching episodes per day, and the amount of time spent feeling nauseous were graded on a 5-point scale. Scores range from 0 (no nausea/distress) to 20 (most nausea/distress).
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Carbidopa | Placebo
Number analyzed (Participants) | 8 | 8
units on a scale | 6.9 (2.2) | 9.7 (2.5)

2. Secondary Outcome: Number of Episodes of Daily Nausea
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: episodes of nausea
Arm/Group | Carbidopa | Placebo
Number analyzed (Participants) | 8 | 8
episodes of nausea | 1.2 (0.8) | 2.0 (1.0)

3. Primary Outcome: 24 Hour Dopamine Levels
Description: Assay of 24 hour dopamine level excretion in urine
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: ug/gCR
Arm/Group | Carbidopa | Placebo
Number analyzed (Participants) | 8 | 8
ug/gCR | 127 (29) | 222 (41)

ADVERSE EVENTS:
Groups:
- Carbidopa: carbidopa
  Carbidopa : The trial will be divided into two consecutive, but independent parts. Phase 1, will address the safety and tolerability of carbidopa in patients with FD using an open-label dose titration phase followed by 4-weeks of open-label treatment. Phase 2, will address the efficacy of carbidopa for the treatment of nausea in patients with FD using a randomized, placebo controlled, double blind, 4-week cross over design.
- Placebo: Placebo
  Placebo : The trial will be divided into two consecutive, but independent parts. Phase 1, will address the safety and tolerability of carbidopa in patients with FD using an open-label dose titration phase followed by 4-weeks of open-label treatment. Phase 2, will address the efficacy of carbidopa for the treatment of nausea in patients with FD using a randomized, placebo controlled, double blind, 4-week cross over design.
Arm/Group | Carbidopa | Placebo
Serious Adverse Events (participants affected / at risk) | 1/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carbidopa (N=12) | Placebo (N=12)
lightheadedness / faint (Nervous system disorders) | 1 (1) | 0 (0) — Patient reported feeling lightheaded and fainted. Blood results indicated patient was anemic and volume depleted, a common feature of FD patients. Patient had a history of dehydration. Patient was hospitalized and recovered without sequelae.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No